CLINICAL TRIAL: NCT00811889
Title: A 52-Week, Multi-center, Double-blind, Randomized, Placebo-controlled Phase IIb Trial to Determine the Effects of Bardoxolone Methyl (RTA 402) on eGFR in Patients With Type 2 Diabetes and Chronic Kidney Disease With an eGFR of 20 - 45 mL/Min/1.73m2
Brief Title: Trial to Determine the Effects of Bardoxolone Methyl on eGFR in Patients With Type 2 Diabetes and Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTA 402-C-0804
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes; Diabetic Nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Bardoxolone Methyl (RTA 402): 75mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl (RTA 402)
- Bardoxolone Methyl (RTA 402): 150mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl (RTA 402)
- Bardoxolone Methyl (RTA 402): 25mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl (RTA 402)

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Placebo
Drug: Bardoxolone Methyl (RTA 402) — Oral, Once Daily
  Arms: Bardoxolone Methyl (RTA 402): 150mg; Bardoxolone Methyl (RTA 402): 25mg; Bardoxolone Methyl (RTA 402): 75mg

SUMMARY:
This study assesses the effects of bardoxolone methyl (RTA 402) in patients with type 2 diabetes and chronic kidney disease.

DETAILED DESCRIPTION:
Bardoxolone methyl (RTA 402) is an Antioxidant Inflammation Modulator (AIM) that is undergoing clinical testing in chronic kidney disease (CKD) and cancer. Bardoxolone methyl and other AIMs inhibit immune-mediated inflammation by restoring redox homeostasis in inflamed tissues by inducing the cytoprotective transcription factor Nrf2. In the diabetic population, adipocytes produce cytokines and mobilize free fatty acids which induce insulin resistance. Resultant hyperglycemia and increased cytokine production induces reactive oxygen and nitrogen species which in turn induce vascular inflammation and endothelial dysfunction. This process causes further activation of NF-kB, creating a vicious cycle of inflammation, vasoconstriction, and ischemia, the end result of which is sclerosis in the kidney and coronary arteries. By inducing Nrf2 and suppressing redox-driven inflammation, we hypothesize that this cycle of inflammation and sclerosis can be abrogated.

Based on Phase IIa data, we hypothesize that bardoxolone methyl will improve renal function through suppression of renal oxidative stress, inflammation and improvement of glomerular filtration. This study was previously posted by Reata Pharmaceuticals. In September 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, at least 18 years of age with known type 2 diabetes, diagnosis of type 2 diabetes should have been made at > 30 years of age (if diabetes developed at a younger age, C-peptide level may be obtained to confirm diagnosis)
2. The average of two eGFR values collected during screening must be within 20 - 45 mL/min/1.73m2, inclusive
3. Patient must be receiving an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 3 months prior to screening, where the dose of the ACE inhibitor or the ARB is considered appropriate for that patient, and has been stable and maintained on that dose for at least 8 weeks prior to the Randomization visit
4. For male and female subjects, agreement to use effective contraception during the entire study period and for at least 2 months after the last dose of study drug, unless documentation of infertility exists
5. Women of child-bearing potential, she must have a negative serum pregnancy test at screening and a negative urine pregnancy test confirmed within 72 hours prior to the first dose of study medication
6. Patient is willing and able to cooperate with all aspects of the protocol
7. Patient is willing and able to give written informed consent for study participation.

Exclusion Criteria:

1. Type 1 (insulin-dependent; juvenile onset) diabetes, or any history of diabetic ketoacidosis
2. Patients with known non-diabetic renal disease or patients with a history of a renal transplant
3. Patients with a Hemoglobin A1c >10% collected at the Screening A visit
4. Cardiovascular disease as follows: Unstable angina pectoris within 3 months prior to study randomization; Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 3 months prior to study randomization; Transient ischemic attack within 3 months of study randomization; Cerebrovascular accident within 3 months of study randomization; Obstructive valvular heart disease or hypertrophic cardiomyopathy; Diagnosis of Class III or IV congestive heart failure at any time
5. Systolic blood pressure (BP) >160 mmHg and diastolic blood pressure > 90 determined by the average of three seated readings taken at least 5 minutes apart, at each of two time-points at least 5 days apart during the screening period
6. QTc Fredericia interval > 450 milliseconds determined by the average of values reported by a central reader from three ECGs taken at the Screening A visit. Each of the three ECGs will be obtained using only equipment provided by the Sponsor, and the ECGs shall be obtained at least ten minutes apart.
7. Second or third degree atrioventricular block not successfully treated with a pacemaker
8. Need for chronic (>2 weeks) immunosuppressive therapy, or need for corticosteroids (excluding intraarticular injections,inhaled or nasal steroids) within 3 months of study randomization
9. Evidence of hepatic or biliary dysfunction including total bilirubin >1.0 mg/dL (>17 micromol/L), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > upper limit of normal (ULN), or alkaline phosphatase >2.0 ULN on ANY screening lab
10. If female, patient is pregnant, nursing or planning a pregnancy
11. Patient has any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the patient while involved in the study or could potentially influence the study outcome
12. Patient has known hypersensitivity to any component of the study drug
13. Patient has undergone a diagnostic or interventional procedure requiring a contrast agent within 30 days prior to randomization
14. Change or dose adjustment in any of the following medications within 8 weeks prior to randomization into the study or anticipated change in dose within 30 days following randomization into the study: ACE inhibitors, angiotensin II receptor blockers.
15. Change or dose adjustment of any other anti-hypertensive, and other anti-diabetic medications within 8 weeks prior to randomization or anticipated change in dose within 30 days following randomization into the study
16. Patient has a current history of drug or alcohol abuse as per the investigator's assessment
17. Patient has participated in another investigational study within 30 days prior to randomization into the study or would concomitantly participate in such a study, or has previously participated in a trial involving bardoxolone methyl.
18. Patient is unable to communicate or cooperate with the investigator due to language problems, poor mental development or impaired cerebral function
19. Patient is unable or unwilling to utilize the daily phone diary to track the date and time they take their study medication
20. Patients on any of the following known hepatotoxic agents: Antioxidant N-acetly-cysteine (Mucomyst, Acetadote, Fluimucil, Parvolex), Niacin (nicotinic acid), Dantrium (dantrolene), Naizide (isoniazid), Normodyne (labetalol), Cylert (pemoline), Felbatol (felbamate), Zyflo (zileuton), Tasmar (tolcapone), or Trovan (trovafloxacin). Patients must have been off the aforementioned medications for a minimum of two weeks prior to randomization
21. Patients who are unable or unwilling to discontinue fenofibrate (Antara, Fenoglide, Lipofen, Lofibra, TriCor, Triglide) during the first three months of study treatment. Patients must have been off fenofibrate for a minimum of two weeks prior to randomization
22. Patients who require more than occasional (once or twice weekly) use of non-steroidal anti-inflammatory agents (NSAIDS)
23. Patients with a history of neoplastic disease (except basal or squamous cell carcinoma of the skin) within 5 years prior to the randomization visit;
24. Patients who have had prior dialysis within three months of randomization and/or have not maintained a stable level of kidney function within three months of randomization per Investigator assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2010-05-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the change in eGFR from baseline in patients with type 2 diabetes and CKD (baseline eGFR = 20 - 45 mL/min/1.73m2) after receiving bardoxolone methyl for 6 months (24 weeks) following randomization | 6 months (24 weeks)
To determine the safety and tolerability of bardoxolone methyl when administered for 12 months (52 weeks)following randomization to type 2 diabetic patients with CKD (eGFR 20 - 45 mL/min/1.73m2). | 1 year (52 weeks)

SECONDARY OUTCOMES:
To quantify the effects of bardoxolone methyl at two different dosing levels relative to placebo on: Hemoglobin A1c, Serum Creatinine, Urine, Intact PTH albumin/creatinine ratio, Serum Phosphorus, Blood Urea Nitrogen, Uric Acid | 6 months (24 weeks) and 1 year (52 weeks)
To determine the change in eGFR from baseline in patients with type 2 diabetes and CKD (baseline eGFR = 20 - 45 mL/min/1.73m2) after receiving bardoxolone methyl for 12 months (52 weeks) following randomization. | 12 months (52 weeks)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Chula Vista, California
  - La Mesa, California
  - Mission Viejo, California
  - Orange, California
  - Riverside, California
  - San Dimas, California
  - Middlebury, Connecticut
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Port Charlotte, Florida
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Baton Rouge, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Flint, Michigan
  - Brooklyn Center, Minnesota
  - Flushing, New York
  - Springfield Gardens, New York
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Roseburg, Oregon
  - Allentown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Salem, Virginia
  - Federal Way, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Pergola PE, Raskin P, Toto RD, Meyer CJ, Huff JW, Grossman EB, Krauth M, Ruiz S, Audhya P, Christ-Schmidt H, Wittes J, Warnock DG; BEAM Study Investigators. Bardoxolone methyl and kidney function in CKD with type 2 diabetes. N Engl J Med. 2011 Jul 28;365(4):327-36. doi: 10.1056/NEJMoa1105351. Epub 2011 Jun 24. PMID 21699484